CLINICAL TRIAL: NCT00589693
Title: A Prospective, Randomized, Double-Blind, Double-Dummy, Multicenter Study to Assess the Safety and Efficacy of Doripenem Compared With Imipenem-Cilastatin in the Treatment of Subjects With Ventilator-Associated Pneumonia
Brief Title: To Compare Safety and Efficacy of Doripenem Versus Imipenem-Cilastatin in Patients With Ventilator-Associated Pneumonia
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Observed lower cure rates and higher mortality rates in one of the treatment groups.
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR014038; DORINOS3008 (Other: Johnson & Johnson Pharmaceutical Research and Development, L.L.C.); 2007-004646-33 (EudraCT Number)
Record Dates: First submitted 2007-12-21; First posted 2008-01-10 (Estimated); Results first posted 2012-07-18 (Estimated); Last update posted 2012-12-28 (Estimated); Status verified 2012-12

CONDITIONS: Ventilator-Associated Pneumonia
Keywords: Ventilator-Associated Pneumonia; Pneumonia, hospital-acquired; Doripenem; Imipenem-cilastatin
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Healthcare-Associated Pneumonia | interventions — Doripenem; Cilastatin, Imipenem Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Doripenem (Experimental): Doripenem from Days 1 to 7 and imipenem-cilastatin placebo from Days 1 to 10
  Interventions: Drug: Doripenem; Drug: Placebo
- Imipenem-Cilastatin (Active Comparator): Imipenem-Cilastatin Days 1 to 10 and doripenem placebo from Days 1 to 7
  Interventions: Drug: Imipenem-Cilastatin; Drug: Placebo

INTERVENTIONS:
Drug: Doripenem — Type=exact number, number=1, unit=g, form=solution for injection, route=intravenously. 1 gram 4-hour infusion of doripenem will be administered every 8 hours for 7 days.
  Arms: Doripenem
Drug: Imipenem-Cilastatin — Type=exact number, number=1, unit=g, form=solution for injection, route=intravenously. 1 gram 1-hour infusion of imipenem-cilastatin will be administered every 8 hours for 10 days.
  Arms: Imipenem-Cilastatin
Drug: Placebo — Form=solution, route=intravenous. Doripenem pacebo will be administered from Days 1 to 7 in imipenem-cilastatin arm and imipenem-cilastatin placebo will be administered in doripenem arm.

SUMMARY:
The purpose of this study is to show that doripenem is as effective as imipenem-cilastatin in the treatment of patients with ventilator-associated pneumonia.

DETAILED DESCRIPTION:
This is a randomized (the study medication is assigned by chance), double-blind (neither physician nor patient knows the treatment that the patient receives), active-controlled (agent that is compared with a study medication to test whether the study medication has a real effect in a clinical study), double-dummy (placebo [inactive substance that is compared with a medication to test whether the medication has a real effect in a clinical study] is administered to maintain the blind when the comparator medication cannot be made identical to the study medication), parallel-group (each group of patients will be treated at the same time), multicenter study to assess the effectiveness and safety of 7 day course of doripenem, compared with 10 day course of imipenem-cilastatin in patients with ventilator-associated pneumonia. This study will consists of 3 phases: (1) a pretreatment phase with a maximum of 24 hours for the screening/baseline visit, (2) a double blind, double dummy, treatment phase of 10 days (Day 1 to Day 10) and an end-of-treatment (EOT) assessment within 24 hours after the last dose of study medication therapy administered on Day 10 or at the time of early withdrawal from study medication, and (3) a post treatment (follow-up) phase consisting of an early follow-up (EFU) visit within 7 to 14 days after the last dose of study medication, and last follow-up (LFU) visit within 28 to 35 days after the last dose of study medication for all patients including those who discontinued study medication early. Two hundred and seventy four patients will be randomly assigned to receive either doripenem or imipenem with placebo of the other medication given simultaneously to maintain the blind (eg, 1 group will receive blinded doripenem from Days 1 to 7 and imipenem placebo Days 1 to 10, other group will receive blinded imipenem Days 1 to 10 and doripenem placebo Days 1 to 7). A sample of secretions from the lower respiratory tract will be obtained by bronchoalveolar lavage (BAL) or mini-BAL within 36 hours prior to administration of study medication from the enrolled patients and sent for culture. Patients, whose baseline BAL or mini-BAL culture results will yield at least 1 qualifying pneumonia pathogen will continue to receive study medication therapy and patients, whose baseline BAL or mini-BAL culture results did not yield at least 1 qualifying pneumonia pathogen will be discontinued from study medication therapy but will remain enroll in the study and will be followed for safety. Safety evaluations including adverse events, clinical laboratory evaluations, vital signs and physical examinations will be monitored throughout the study period. The total duration of an individual patient's participation in the study will be approximately 5 to 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have new or worsening radiographic infiltrates consistent with ventilator-associated pneumonia that was not related to cardiac or other disease processes
* Have at least 1 of the following: fever (core body temperature greater than 39.0°C); hypothermia (core body temperature of less than 35.0°C); leukocytosis (increased WBC count); and leukopenia (decreased WBC count)
* Have developed ventilator-associated pneumonia and have been on mechanical ventilation for more than or equal to 48 hours and on mechanical ventilation at the time that study medication is assigned
* Have been hospitalized or been in a chronic care facility for consecutive 5 days or more within the last 90 days
* Have a baseline Clinical Pulmonary Infection Score (CPIS) more than or equal to 6 and an Acute Physiology and Chronic Health Evaluation (APACHE) II score more than 8 and less than 35

Exclusion Criteria:

* Have received antibiotics for this episode of ventilator-associated pneumonia for more than 24 hours before study medication administration
* Known presence at baseline of only methicillin-resistant Staphylococcus aureus or Stenotrophomonas infection
* Acute respiratory distress syndrome
* Has any of the following conditions: chest trauma with severe lung bruising or loss of stability of the thoracic cage following a fracture of the sternum, ribs, or both, increased amounts of fluid in the lung cavities requiring drainage or pus in the cavity
* Has active seizure disorder within the last 2 years or brain injury such that imipenem cilastatin would not be administered to the patient in usual practice
* Has lung cancer within the last 2 years, chronic bronchitis with an increase in severity within the last 30 days, chronic enlargement of the bronchi or bronchioles related to inflammatory disease or obstruction, lung abscess(s), anatomical bronchial obstruction, respiratory tuberculosis on treatment, suspected atypical pneumonia, chemical pneumonitis, cystic fibrosis, congestive heart failure, severe burns to greater than 15% of the body, evidence of severe and chronic liver disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Actual)
Dates: Start 2008-04; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (100):
- United States (17):
  - Jonesboro, Arkansas
  - Newark, Delaware
  - Washington D.C., District of Columbia
  - Jacksonville, Florida
  - Moline, Illinois
  - Hazard, Kentucky
  - Biddeford, Maine
  - Baltimore, Maryland
  - Detroit, Michigan
  - Butte, Montana
  - Buffalo, New York
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Oklahoma City, Oklahoma
  - Nashville, Tennessee
  - Houston, Texas
  - Milwaukee, Wisconsin
- Argentina (6):
  - Buenos Aires
  - Córdoba
  - Entre Ríos
  - Monte Grande
  - Rio Negro
  - Rosario
- Australia (5):
  - Adelaide
  - Box Hill
  - Clayton
  - Melbourne
  - Parkville
- Belgium (2):
  - Brussels
  - Ghent
- Brazil (8):
  - Belo Horizonte
  - Curitiba
  - Fortaleza
  - Porto Alegre
  - Rio de Janeiro
  - Santo André
  - São José do Rio Preto
  - São Paulo
- Canada (3):
  - Halifax, Nova Scotia
  - Ottawa, Ontario
  - Greenfield Park, Quebec
- France (5):
  - Argenteuil
  - Limoges
  - Paris
  - Pierre-Bénite
  - Tours
- Germany (6):
  - Dresden
  - Halle
  - Homburg/Saar
  - Lübeck
  - Mannheim
  - Ulm
- Guatemala (3):
  - Cuilapa
  - Escuintla Escuintla
  - Guatemala City
- Hungary (3):
  - Budapest
  - Budapest Na
  - Székesfehérvár
- India (5):
  - Bangalore
  - Coimbatore
  - Ludhiana
  - New Delhi
  - Pune
- Israel (3):
  - Afula
  - Petah Tikva
  - Ramat Gan
- Mexico (5):
  - Chihuahua City
  - Guadalajara
  - Monterrey
  - San Luis Potosí City
  - Zapopan
- Philippines (2):
  - Manila
  - Quezon City
- Portugal (2):
  - Lisbon
  - Porto
- Romania (3):
  - Brasov
  - Târgu Mureş
  - Timișoara
- Russia (5):
  - Moscow
  - Saint Petersburg
  - Saratov
  - Smolensk
  - Yaroslavl
- Spain (5):
  - Barcelona
  - L'Hospitalet de Llobregat
  - Las Palmas de Gran Canaria
  - Madrid
  - Tarragona
- Thailand (3):
  - Chiang Mai
  - Khon Kaen
  - Nakhonratchasima
- Turkey (Türkiye) (6):
  - Adana
  - Ankara
  - Istanbul
  - Kayseri
  - Samsun
  - Trabzon
- Ukraine (3):
  - Kharkiv
  - Kiev
  - Odesa

REFERENCES:
- [Derived] Kollef MH, Chastre J, Clavel M, Restrepo MI, Michiels B, Kaniga K, Cirillo I, Kimko H, Redman R. A randomized trial of 7-day doripenem versus 10-day imipenem-cilastatin for ventilator-associated pneumonia. Crit Care. 2012 Nov 13;16(6):R218. doi: 10.1186/cc11862. PMID 23148736

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 274 enrolled patients were randomnly assigned to the 127 study centers. 524 patients were to be enrolled, however as the study was terminated early only 274 patients were actually enrolled.
Pre-assignment Details: Out of 274 randomized patients, 41 patients were excluded (as their sites were GCP Non-Compliant) and 6 patients were not treated. Treated patients=227 (115 doripenem and 112 imipenem-cilastatin).
Groups:
- Doripenem: 1 g 4-hour infusion intravenously every 8 hour for 7 days
- Imipenem-cilastatin: 1 g 1-hour infusion intravenously every 8 hour for 10 days
Period: Overall Study
Arm/Group | Doripenem | Imipenem-cilastatin
Started | 115 | 112
Completed | 71 | 83
Not Completed | 44 | 29
Not completed — randomized in error | 12 | 6
Not completed — Adverse Event | 4 | 4
Not completed — Death | 26 | 16
Not completed — Lack of Efficacy | 0 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 0 | 1
Not completed — Protocol Violation | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Doripenem | Imipenem-cilastatin | Total
Number analyzed (Participants) | 115 | 112 | 227
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1
  Between 18 and 65 years | 72 | 72 | 144
  >=65 years | 43 | 39 | 82
Age Continuous [Mean (Standard Deviation); unit: years] | 57.5 (16.53) | 54.6 (18.46) | 56.1 (17.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 37 | 80
  Male | 72 | 75 | 147
Region Enroll [Number; unit: participants]
  EUROPE | 69 | 71 | 140
  NORTH AMERICA | 16 | 12 | 28
  REST OF WORLD | 9 | 6 | 15
  SOUTH AMERICA | 21 | 23 | 44

OUTCOME MEASURES:

1. Primary Outcome: Clinical Cure Rate at the End-of-treatment (EOT) Visit
Description: The number of patients who achieved clinical cure at the EOT visit on Day 10. The patient's were classified as clinical cure if they had resolution of signs and symptoms and objective findings of pneumonia to such an extent that no further antimicrobial therapy was necessary.
Time Frame: End-of-treatment (Day 10 or Day 11)
Population: Microbiological Intent-to-Treat (MITT) - subset of all ITT (all randomized patients who received at least a partial dose of study medication) patients who had at least 1 qualifying pneumonia pathogen.
Measure: Number; unit: Participants
Arm/Group | Doripenem | Imipenem-cilastatin
Number analyzed (Participants) | 79 | 88
Participants | 36 | 50
Statistical Analysis 1: Comparison: Doripenem vs Imipenem-cilastatin; Null Hypothesis: The clinical cure rate of doripenem assessed at the EOT visit is more than 15% inferior to that of imipenem-cilastatin; Test type: Non-Inferiority or Equivalence — Noninferiority will be established if the lower limit of the 2-sided 95% Confidence Interval (CI) of the difference in clinical cure rate (doripenem minus imipenem-cilastatin) is greater than 15%; Normal approximation of 2 proportions; Difference of 2 binomial proportions = -11.2, 95% CI 2-sided [-26.3 to 3.8]

2. Secondary Outcome: Clinical Cure Rate at the End-of-treatment (EOT) Visit in Patients From Whom a Qualifying P. Aeruginosa Was Isolated at Baseline
Description: The clinical cure rate at the EOT visit in patients, whose bronchoalveolar lavage (BAL) or mini-BAL culture results yielded qualifying pneumonia pathogen P. aeruginosa at baseline.
Time Frame: End-of-treatment (Day 10 or Day 11)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Doripenem | Imipenem-cilastatin
Number analyzed (Participants) | 17 | 10
Participants | 7 | 6
Statistical Analysis 1: Comparison: Doripenem vs Imipenem-cilastatin; Test type: Superiority or Other; Normal approximation of 2 proportions; Difference of 2 binomial proportions = -18.8, 95% CI 2-sided [-57.2 to 19.5]

3. Secondary Outcome: Clinical Cure Rate at the End-of-treatment (EOT) Visit in Patients From Whom at Least 1 of the Gram-negative Qualifying Pneumonia Pathogens (Enterobacteriaceae, P. Aeruginosa, and Acinetobacter Spp) Was Isolated at Baseline
Description: The clinical cure rate at the EOT visit in patients whose BAL or mini-BAL culture results yielded at least 1 of the following Gram-negative qualifying pneumonia pathogens was isolated at baseline: any Enterobacteriaceae, P. aeruginosa, and Acinetobacter Spp.
Time Frame: End-of-treatment (Day 10 or Day 11)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Doripenem | Imipenem-cilastatin
Number analyzed (Participants) | 65 | 62
Participants | 32 | 34
Statistical Analysis 1: Comparison: Doripenem vs Imipenem-cilastatin; Test type: Superiority or Other; Normal approximation of 2 proportions; Difference of 2 binomial proportions = -5.6, 95% CI 2-sided [-23.0 to 11.7]

4. Secondary Outcome: Number of Patients Who Had Emergence of P. Aeruginosa Resistance
Description: Number of patients who had P. aeruginosa isolates with a 4 fold or greater increase in minimum inhibitory concentration (MIC) at anytime during the study (after the study medication is received) from baseline
Time Frame: Up to 6 weeks
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Doripenem | Imipenem-cilastatin
Number analyzed (Participants) | 19 | 15
Participants | 3 | 6
Statistical Analysis 1: Comparison: Doripenem vs Imipenem-cilastatin; Test type: Superiority or Other; p = 0.14, Fisher Exact

5. Secondary Outcome: 28-day All-cause Mortality Rate
Description: Number of deaths which occured up to 28 days of the study period due to all causes
Time Frame: Up to 28 days
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Doripenem | Imipenem-cilastatin
Number analyzed (Participants) | 79 | 88
Participants | 17 | 13
Statistical Analysis 1: Comparison: Doripenem vs Imipenem-cilastatin; Test type: Superiority or Other; Normal approximation of 2 proportions; Difference of 2 binomial proportions = 6.7, 95% CI 2-sided [-5.0 to 18.5]

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: Only patients who had at least one of the treatment related adverse events (AEs) was listed in the other (non Serious) AE table and was included as the total number of patients with Non-Serious Adverse Events.
Arm/Group | Doripenem | Imipenem-cilastatin
Serious Adverse Events (participants affected / at risk) | 55/115 | 45/112
Other Adverse Events (participants affected / at risk) | 82/115 | 80/112
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Doripenem (N=115) | Imipenem-cilastatin (N=112)
Sepsis (Infections and infestations) | 8 | 3
Septic shock (Infections and infestations) | 6 | 6
Pneumonia (Infections and infestations) | 5 | 3
Device related sepsis (Infections and infestations) | 3 | 2
Urinary tract infection (Infections and infestations) | 3 | 1
Empyema (Infections and infestations) | 2 | 0
Abscess (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 2
Central nervous system infection (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Infected skin ulcer (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 1 | 1
Pneumonia bacterial (Infections and infestations) | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 0
Staphylococcal skin infection (Infections and infestations) | 1 | 0
Superinfection (Infections and infestations) | 1 | 0
Abdominal abscess (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 0 | 1
Fungal infection (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 0 | 1
Mediastinitis (Infections and infestations) | 0 | 2
Meningitis (Infections and infestations) | 0 | 1
Pneumonia klebsiella (Infections and infestations) | 0 | 1
Postoperative wound infection (Infections and infestations) | 0 | 1
Pulmonary sepsis (Infections and infestations) | 0 | 2
Tracheobronchitis (Infections and infestations) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Pleural disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 3 | 6
Cardiac failure (Cardiac disorders) | 2 | 3
Atrial fibrillation (Cardiac disorders) | 1 | 0
Bradyarrhythmia (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 2
Renal failure (Renal and urinary disorders) | 5 | 1
Renal failure acute (Renal and urinary disorders) | 2 | 2
Acute prerenal failure (Renal and urinary disorders) | 1 | 0
Renal tubular acidosis (Renal and urinary disorders) | 0 | 1
Brain oedema (Nervous system disorders) | 3 | 4
Intracranial pressure increased (Nervous system disorders) | 2 | 1
Brain stem syndrome (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Nervous system disorder (Nervous system disorders) | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Hydrocephalus (Nervous system disorders) | 0 | 1
Subdural hygroma (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Traumatic brain injury (Injury, poisoning and procedural complications) | 3 | 0
Fat embolism (Injury, poisoning and procedural complications) | 1 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 1 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 | 1
Extradural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Spinal cord injury cervical (Injury, poisoning and procedural complications) | 0 | 1
Duodenal perforation (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Pancreatic necrosis (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Peritonitis (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1
Ileus paralytic (Gastrointestinal disorders) | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Multi-organ failure (General disorders) | 2 | 3
Treatment failure (General disorders) | 2 | 0
Impaired healing (General disorders) | 0 | 1
Circulatory collapse (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Hypovolaemic shock (Vascular disorders) | 1 | 0
Intra-abdominal haemorrhage (Vascular disorders) | 1 | 0
Shock (Vascular disorders) | 1 | 2
Haemorrhage (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 3
Jugular vein thrombosis (Vascular disorders) | 0 | 1
Thrombosis (Vascular disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Diabetes insipidus (Endocrine disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 1
Hypersensitivity (Immune system disorders) | 1 | 0
Troponin increased (Investigations) | 1 | 0
Metastases to pleura (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Doripenem (N=115) | Imipenem-cilastatin (N=112)
Diarrhoea (Gastrointestinal disorders) | 11 | 12
Constipation (Gastrointestinal disorders) | 9 | 11
Vomiting (Gastrointestinal disorders) | 6 | 6
Nausea (Gastrointestinal disorders) | 5 | 7
Depression (Psychiatric disorders) | 14 | 8
Agitation (Psychiatric disorders) | 11 | 7
Insomnia (Psychiatric disorders) | 8 | 8
Anxiety (Psychiatric disorders) | 2 | 6
Anaemia (Blood and lymphatic system disorders) | 26 | 25
Hypokalaemia (Metabolism and nutrition disorders) | 12 | 12
Hyperkalaemia (Metabolism and nutrition disorders) | 6 | 6
Hypernatraemia (Metabolism and nutrition disorders) | 5 | 7
Hyponatraemia (Metabolism and nutrition disorders) | 5 | 10
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 | 7
Urinary tract infection (Infections and infestations) | 13 | 16
Pneumonia (Infections and infestations) | 6 | 9
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 14 | 11
Hypotension (Vascular disorders) | 11 | 8
Hypertension (Vascular disorders) | 2 | 6
Atrial fibrillation (Cardiac disorders) | 9 | 8
Bradycardia (Cardiac disorders) | 3 | 6
Pyrexia (General disorders) | 11 | 10
Renal impairment (Renal and urinary disorders) | 6 | 4
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 4 | 6

LIMITATIONS AND CAVEATS:
41 patients (21 doripenem, 20 imipenem-cilastatin) were enrolled at 5 sites that were found to be Good Clinical Practice non-compliant and were excluded from the primary efficacy and safety analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days